CLINICAL TRIAL: NCT00996164
Title: A Twenty-four Week, Randomized, Double-blind, Placebo Controlled, Safety and Efficacy Trial of Flibanserin (100 Milligrams) Administered Orally Once Daily in Premenopausal Women With Hypoactive Sexual Desire Disorder in the United States
Brief Title: Fixed 100 mg Every Evening of Flibanserin vs Placebo in Premenopausal Women With Hypoactive Sexual Desire Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sprout Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 511.147
Record Dates: First submitted 2009-10-15; First posted 2009-10-16 (Estimated); Results first posted 2014-05-19 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-04

CONDITIONS: Sexual Dysfunctions, Psychological
MeSH Terms: conditions — Sexual Dysfunctions, Psychological | interventions — flibanserin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- flibanserin 100 mg (Experimental): flibanserin 100mg po qd
  Interventions: Drug: Flibanserin
- Placebo (Placebo Comparator): placebo 1 tab po qd
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Flibanserin — patients will be randomized to flibanserin or placebo in a double-blind manner
  Arms: flibanserin 100 mg
Drug: Placebo — patients will be randomized to flibanserin or placebo in a double-blind manner
  Arms: Placebo

SUMMARY:
The object of this trial is to assess the safety and efficacy of a 24 week course of flibanserin for the treatment of hypoactive sexual desire disorder in premenopausal women.

ELIGIBILITY:
Inclusion criteria:

1. Premenopausal women who are 18 years old and older
2. Primary diagnosis of hypoactive sexual desire disorder, generalized acquired type according to Diagnostic and Statistical Manual of Mental Disorder, Fourth Edition, Text Revision, at least 24 weeks in duration.
3. Stable, monogamous heterosexual relationship for at least one year.
4. Willing to discuss sexual issues.
5. Willing to engage in sexual activity at least once a month
6. Normal pap smear
7. Must use medically acceptable method of contraception
8. Able to comply with daily use of a handheld entry device

Exclusion criteria:

1. Patients who have taken any medication in the protocol List of Prohibited Medications within 30 days before the screening visit.
2. Patients who meet Diagnostic and Statistical Manual of Mental Disorder, Fourth Edition, Text Revision for: Sexual aversion disorder, substance induced sexual dysfunction, Dyspareunia, vaginismus, gender identity disorder, paraphilia, sexual dysfunction do to a general medical condition.
3. Partner with inadequately treated organic or psychosexual dysfunction
4. History of Major Depressive Disorder within six months prior to the screening visit or history of suicidal behavior.
5. Sexual function impaired by psychiatric disorder
6. Sexual function impaired by gynecological disorder
7. Major life stress that could impair sexual function
8. Substance abuse

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1090 (Actual)
Dates: Start 2009-10; Primary Completion 2010-12 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (75):
- United States (75):
  - 511.147.01074 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 511.147.01046 Boehringer Ingelheim Investigational Site, Huntsville, Alabama
  - 511.147.01042 Boehringer Ingelheim Investigational Site, Mobile, Alabama
  - 511.147.01025 Boehringer Ingelheim Investigational Site, Phoenix, Arizona
  - 511.147.01073 Boehringer Ingelheim Investigational Site, Phoenix, Arizona
  - 511.147.01030 Boehringer Ingelheim Investigational Site, Encinitas, California
  - 511.147.01028 Boehringer Ingelheim Investigational Site, Fair Oaks, California
  - 511.147.01037 Boehringer Ingelheim Investigational Site, Irvine, California
  - 511.147.01022 Boehringer Ingelheim Investigational Site, Sacramento, California
  - 511.147.01035 Boehringer Ingelheim Investigational Site, San Diego, California
  - 511.147.01052 Boehringer Ingelheim Investigational Site, San Diego, California
  - 511.147.01016 Boehringer Ingelheim Investigational Site, Torrance, California
  - 511.147.01021 Boehringer Ingelheim Investigational Site, Vista, California
  - 511.147.01051 Boehringer Ingelheim Investigational Site, Westlake Village, California
  - 511.147.01071 Boehringer Ingelheim Investigational Site, Denver, Colorado
  - 511.147.01053 Boehringer Ingelheim Investigational Site, Farmington, Connecticut
  - 511.147.01015 Boehringer Ingelheim Investigational Site, Groton, Connecticut
  - 511.147.01041 Boehringer Ingelheim Investigational Site, New Britain, Connecticut
  - 511.147.01064 Boehringer Ingelheim Investigational Site, Newark, Delaware
  - 511.147.01062 Boehringer Ingelheim Investigational Site, Washington D.C., District of Columbia
  - 511.147.01003 Boehringer Ingelheim Investigational Site, Boynton Beach, Florida
  - 511.147.01056 Boehringer Ingelheim Investigational Site, Clearwater, Florida
  - 511.147.01065 Boehringer Ingelheim Investigational Site, Daytona Beach, Florida
  - 511.147.01020 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 511.147.01024 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 511.147.01070 Boehringer Ingelheim Investigational Site, New Port Richey, Florida
  - 511.147.01043 Boehringer Ingelheim Investigational Site, Orlando, Florida
  - 511.147.01019 Boehringer Ingelheim Investigational Site, St. Petersburg, Florida
  - 511.147.01061 Boehringer Ingelheim Investigational Site, Tampa, Florida
  - 511.147.01066 Boehringer Ingelheim Investigational Site, Tampa, Florida
  - 511.147.01001 Boehringer Ingelheim Investigational Site, West Palm Beach, Florida
  - 511.147.01002 Boehringer Ingelheim Investigational Site, West Palm Beach, Florida
  - 511.147.01009 Boehringer Ingelheim Investigational Site, Atlanta, Georgia
  - 511.147.01023 Boehringer Ingelheim Investigational Site, Atlanta, Georgia
  - 511.147.01008 Boehringer Ingelheim Investigational Site, Sandy Springs, Georgia
  - 511.147.01044 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 511.147.01034 Boehringer Ingelheim Investigational Site, Indianapolis, Indiana
  - 511.147.01067 Boehringer Ingelheim Investigational Site, Lafayette, Louisiana
  - 511.147.01013 Boehringer Ingelheim Investigational Site, Baltimore, Maryland
  - 511.147.01031 Boehringer Ingelheim Investigational Site, Bingham Farms, Michigan
  - 511.147.01006 Boehringer Ingelheim Investigational Site, St Louis, Missouri
  - 511.147.01014 Boehringer Ingelheim Investigational Site, Billings, Montana
  - 511.147.01060 Boehringer Ingelheim Investigational Site, Omaha, Nebraska
  - 511.147.01057 Boehringer Ingelheim Investigational Site, Las Vegas, Nevada
  - 511.147.01039 Boehringer Ingelheim Investigational Site, Moorestown, New Jersey
  - 511.147.01017 Boehringer Ingelheim Investigational Site, Endwell, New York
  - 511.147.01047 Boehringer Ingelheim Investigational Site, New Bern, North Carolina
  - 511.147.01027 Boehringer Ingelheim Investigational Site, Winston-Salem, North Carolina
  - 511.147.01033 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 511.147.01004 Boehringer Ingelheim Investigational Site, Cleveland, Ohio
  - 511.147.01050 Boehringer Ingelheim Investigational Site, Columbus, Ohio
  - 511.147.01059 Boehringer Ingelheim Investigational Site, Columbus, Ohio
  - 511.147.01058 Boehringer Ingelheim Investigational Site, Dayton, Ohio
  - 511.147.01072 Boehringer Ingelheim Investigational Site, Oklahoma City, Oklahoma
  - 511.147.01007 Boehringer Ingelheim Investigational Site, Eugene, Oregon
  - 511.147.01055 Boehringer Ingelheim Investigational Site, Pittsburgh, Pennsylvania
  - 511.147.01048 Boehringer Ingelheim Investigational Site, Columbia, South Carolina
  - 511.147.01068 Boehringer Ingelheim Investigational Site, Mt. Pleasant, South Carolina
  - 511.147.01063 Boehringer Ingelheim Investigational Site, Knoxville, Tennessee
  - 511.147.01010 Boehringer Ingelheim Investigational Site, Nashville, Tennessee
  - 511.147.01036 Boehringer Ingelheim Investigational Site, Nashville, Tennessee
  - 511.147.01018 Boehringer Ingelheim Investigational Site, Corpus Christi, Texas
  - 511.147.01032 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 511.147.01011 Boehringer Ingelheim Investigational Site, Katy, Texas
  - 511.147.01012 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 511.147.01026 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 511.147.01005 Boehringer Ingelheim Investigational Site, Salt Lake City, Utah
  - 511.147.01069 Boehringer Ingelheim Investigational Site, Sandy City, Utah
  - 511.147.01040 Boehringer Ingelheim Investigational Site, Norfolk, Virginia
  - 511.147.01049 Boehringer Ingelheim Investigational Site, Norfolk, Virginia
  - 511.147.01029 Boehringer Ingelheim Investigational Site, Richmond, Virginia
  - 511.147.01075 Boehringer Ingelheim Investigational Site, Richmond, Virginia
  - 511.147.01054 Boehringer Ingelheim Investigational Site, Renton, Washington
  - 511.147.01045 Boehringer Ingelheim Investigational Site, Spokane, Washington
  - 511.147.01038 Boehringer Ingelheim Investigational Site, Tacoma, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Flibanserin 100 mg | Placebo
Started | 543 | 547
Completed | 408 | 446
Not Completed | 135 | 101

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Flibanserin 100 mg | Placebo | Total
Number analyzed (Participants) | 543 | 547 | 1090
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 543 | 547 | 1090
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.5 (7.8) | 36.6 (8.0) | 36.5 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 543 | 547 | 1090
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 543 | 547 | 1090

OUTCOME MEASURES:

1. Primary Outcome: The Change From Baseline to Week 24 in the Score of the Female Sexual Function Index Desire Domain.
Description: The FSFI is a self-administered questionnaire for assessing key dimensions of sexual function in women. The scale consists of 19 items assessing sexual function over the past 4 weeks and yields scores in 6 domains: desire, arousal, lubrication, orgasm, satisfaction, and pain. The 2 items in the desire domain are scored from '1' to '5'. The raw scores of the 2 items are added together and then multiplied by the domain factor of 0.6. Thus, the score of the desire domain ranges from 1.2 to 6.0. The higher the score on the desire domain, the higher the level of reported sexual desire.
Time Frame: 24 weeks
Population: The Full Analysis Set (FAS) consisted of those patients who were randomized to a treatment group, received at least one dose of study medication, and had at least one on-treatment efficacy assessment. The treated set was analyzed for safety. The FAS was analyzed for efficacy.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Flibanserin 100 mg | Placebo
Number analyzed (Participants) | 506 | 525
units on a scale | 1.0 (0.1) | 0.7 (0.1)

2. Primary Outcome: Change From Baseline in the SSE Count From Baseline to 24 Weeks
Description: The change from baseline in the number of Satisfying Sexual Events (SSEs) as measured by the eDiary. The SSEs will be standardized to a 28-day period according to the below formula:
  Total monthly events = 28 x (sum of the number of events) / (sum of number of days entered).
  "Satisfying" means gratifying, fulfilling, satisfactory, and/or successful for the patient. The partner's satisfaction is not the subject of this question.
  An eDiary was used by the patients to record information about sexual events. Patients were instructed to complete the eDiary every morning. When completing an eDiary entry, patients answered questions regarding their sexual events since their last eDiary entry. If patients missed or were late with their eDiary entry, they entered information about their sexual events covering a maximum time period of the past 7 days; however, they did not enter any information beyond the last entry.
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: SSEs
Arm/Group | Flibanserin 100 mg | Placebo
Number analyzed (Participants) | 500 | 521
SSEs | 2.5 (4.6) | 1.5 (4.5)

ADVERSE EVENTS:
Arm/Group | Flibanserin 100 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 4/543 | 2/547
Other Adverse Events (participants affected / at risk) | 237/543 | 68/547
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flibanserin 100 mg (N=543) | Placebo (N=547)
suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
biliary dyskinesia (Hepatobiliary disorders) | 1 (1) | 0 (0)
cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flibanserin 100 mg (N=543) | Placebo (N=547)
somnolence (Nervous system disorders) | 78 (81) | 19 (19)
dizziness (Nervous system disorders) | 56 (62) | 6 (6)
nausea (Gastrointestinal disorders) | 41 (44) | 12 (12)
fatigue (Nervous system disorders) | 32 (32) | 18 (18)
upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 30 (31) | 13 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No